CLINICAL TRIAL: NCT04068207
Title: The Efficacy and Safety of Oral Minocycline in the Treatment of Retinitis Pigmentosa: An Open-label Clinical Trial
Brief Title: Minocycline Treatment in Retinitis Pigmentosa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Dan Liang, Lab of ocular immunology in Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5010-MINO-RP
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-04

CONDITIONS: Retinitis Pigmentosa; Inherited Retinal Dystrophy; Retina Disorder
Keywords: Retinitis Pigmentosa; Minocycline; ERG; Inherited Retinal Dystrophy; Retinal Degenerative Disease
MeSH Terms: conditions — Retinitis Pigmentosa; Retinal Diseases; cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Minocycline (Experimental): Tablets Minocycline 100mg po per day for 12 months
  Interventions: Drug: Minocycline

INTERVENTIONS:
Drug: Minocycline — Tab. Minocycline 100mg po per day for 12 months
  Other Names: Minocin; Minocyclinum; Minocyclin

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of oral minocycline (100mg/d), administered for 6 months, for the treatment of patients with retinitis pigments(RP).

DETAILED DESCRIPTION:
Retinitis Pigmentosa (RP)is a sort of inherited blinding disorders and no effective or safe treatment are widely applied for it. The worldwide prevalence of RP is estimated to be 1/5000. RP is characterized by degeneration of peripheral rod photoreceptor(PR) and associated retinal pigment epithelium(RPE) cells. Nyctalopia and visual field constriction are common symptoms. Cone degeneration and associated loss of central vision are typically followed later.

Minocycline, a secord-generation, semi-synthetic tetracycline antibiotic, is a highly lipophilic molecule and can easily pass through the blood-brain barrier. Several animal experiments and clinical trials have reported that minocycline exert anti-apoptotic, anti-inflammatory and antioxidant effects in treating neurodegenerative diseases.

We propose to test the effect and safety of oral minocycline for retinitis pigmentosa.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Retinitis Pigmentosa: nyctalopia, visual field constriction and loss of central vision; degeneration of peripheral rod photoreceptor and retinal pigment epithelium cells.
* Age from 18 to 60 years old.
* BCVA >20/100(0.2) at least in one eye.
* Full-field cone electroretinogram amplitude to 30-Hz flashes >0uV at least in one eye.
* Written informed consent is provided.

Exclusion Criteria:

* Glucocortticoids or tetracycline were used within 3 months.
* Vitamin A, DHA and other neurotrophic drugs were used within 3 months.
* Other ocular diseases or fundus diseases except cataract: glaucoma, diabetic retinopathy, retinal detachment.
* Tetracycline or minocycline allergy or intolerance.
* Renal or hepatic insufficiency.
* History of thyroid neoplasm.
* History of idiopathic intracranial hypertension.
* Pregnant or lactating females.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2019-08-25 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
change of full-field cone electroretinogram amplitude to 30-Hz flashes | 12 months， 24 weeks
  increase of full-field cone electroretinogram amplitude to 30-Hz flashes

SECONDARY OUTCOMES:
change of visual field area | 12 months， 24 weeks
  HFA30-2 and HFA60-4
Best Corrected Visual Acuity | 12 months， 24 weeks
  increase of BCVA
other ERG indexes | 12 months， 24 weeks
  ERG indexes
color vision | 12 months， 24 weeks
  Farnsworth-Munsell 100-hue test (FM-100)
Contrast sensitivity | 12 months， 24 weeks
  Functional Acuity Contrast Test (FACT)
central foveal thickness | 12 months， 24 weeks
  central foveal thickness via OCT

CONTACTS AND LOCATIONS:
Overall Officials: Dan Liang, MD, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Chen Y, Pan Y, Xie Y, Shi Y, Lu Y, Xia Y, Su W, Chen X, Li Z, Wang M, Miao S, Yang Y, Jin C, Luo G, Long S, Xiao H, Huang C, Zhang J, Liang D. Efficacy and safety of minocycline in retinitis pigmentosa: a prospective, open-label, single-arm trial. Signal Transduct Target Ther. 2024 Dec 4;9(1):339. doi: 10.1038/s41392-024-02037-2. PMID 39627217